CLINICAL TRIAL: NCT02973113
Title: Phase I Study Combining Nivolumab With Epstein Barr Virus Specific T Cells (EBVSTS) in Relapsed/Refractory EBV Positive Lymphoma Patients (PREVALE)
Brief Title: Nivolumab With Epstein Barr Virus Specific T Cells (EBVSTS), Relapsed/Refractory EBV Positive Lymphoma (PREVALE)
Acronym: PREVALE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Director CAGT, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-39090 PREVALE; PREVALE (Other: Baylor College of Medicine)
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: NonHodgkin Lymphoma; Lymphoproliferative Disorders; EBV Related Lymphoma; EBV-Related PTLD; Hodgkin Lymphoma; EBV Related Non-Hodgkin's Lymphoma; EBV Related Hodgkin's Lymphoma
Keywords: Nivolumab; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Lymphoproliferative Disorders; EBV-specific T Cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EBVST Cells + Nivolumab (Experimental): PD1 inhibitor - nivolumab 3 mg/kg (max dose: 240 mg) Q 2 weeks for total 4 doses and repeat a day prior to each EBVST infusion.
  EBVST- 1 x 10^8/m2 at days +1 and +15. PD1 inhibitor - nivolumab 3 mg/kg (max dose: 240 mg) Q 2 weeks for total 4 doses and repeat a day prior to each EBVST infusion.
  Can receive up to 3 additional infusions of EBVSTs with a single dose of nivolumab at 6-12 week intervals starting at least 6 weeks after the second infusion if stable disease or a partial response at Week 8 evaluation
  Interventions: Biological: EBVST Cells; Biological: Nivolumab

INTERVENTIONS:
Biological: EBVST Cells — EBVST cells in an expected volume of 10-20cc will be given by intravenous injection over 2-10 minutes through either a peripheral or a central line.
  Other Names: EBV-specific T Cells
Biological: Nivolumab — Nivolumab 3mg/kg (max dose: 240 mg) will be administered as an intravenous infusion over 60 minutes.
  Other Names: Opdivo

SUMMARY:
Subjects have a type of a lymph node cancer called Non-Hodgkin's Lymphoma (NHL) or lymphoproliferative disease (LPD), which affects their immunity, blood production, and can involve multiple other organs in the body. Their disease has come back or has not gone away after treatment. The experimental treatment plan consists of an antibody therapy called "Nivolumab" that helps the subjects' T-cells control the tumor, and special immune system cells called EBV-specific cytotoxic T lymphocytes, also a new therapy whose side effects are well studied.

Some patients with NHL or LPD are infected with the virus that causes infectious mononucleosis (called Epstein-Barr virus, or EBV) before or at the time of their diagnosis. The cancer cells that are infected by EBV are able to hide from the body's immune system and escape destruction. Investigators want to see if special white blood cells, called T cells, that have been trained to kill cells infected by EBV can survive in the blood and affect the tumor.

Investigators have used this sort of therapy to treat a different type of cancer that occurs after bone marrow or solid organ transplant called post-transplant lymphoma with good success. These cells are called EBV-specific cytotoxic T-lymphocytes (EBVSTs), and are effective in treating these diseases. These EBVSTs are experimental and not yet approved by the Food and Drug Administration (FDA).

Sometimes it is not possible to grow these cells; or they may not last very long in the body after being given into the vein thereby having only limited time to fight the tumor. With this study, investigators aim to increase the duration of time that the T cells can last in the body and can effectively fight the cancer by using nivolumab. Nivolumab is FDA approved for treatment of other kinds of cancer like lung cancer and a skin cancer called Melanoma.

The purpose of this study is to find out if EBVST cells in combination with nivolumab are safe, to learn what the side effects are, and to see whether this therapy may help patients with EBV related lymphoma or LPD.

DETAILED DESCRIPTION:
The investigators will draw blood from the subject to make EBV-specific cytotoxic T-lymphocytes (EBVSTs) in the lab. Investigators will make the cells by first growing a special type of cells called dendritic cells (DCs) or monocytes to stimulate the T cells. Then they will add specially produced mixtures of proteins that included the LMP, EBNA1, and BARF proteins. These are used to stimulate T cells. As the T cells grow, investigators add some of the subject's cells expressing these proteins to stimulate them. They also add a cell called K562 that has had new genes put inside it so it expresses proteins that stimulate the immune system to encourage the T cells to grow. This stimulation trains the EBVSTs to kill cells with EBV proteins on their surface. These cells will be grown and frozen.

The cells grown in the lab will be thawed and injected into the subject's vein over 2-10 minutes. Initially, one dose of the drug nivolumab is given one day before the EBVST cells are infused (on day 0) and then every 2 weeks for a total of four doses of nivolumab. Subjects will receive two infusions of the EBVST cells. The first infusion will be given on Day 1 and a second infusion of T cells on Day 15.

If eligible, subjects may receive up to three additional doses of the T cells 6-12 weeks apart and each additional T cell infusion would be preceded by one dose of nivolumab a day prior.

Subjects will have medical and blood tests at predetermined time points. Investigators will follow subjects closely after treatment for any side effects for at least for 1 year after the subject's last infusion.

ELIGIBILITY:
Inclusion Criteria:

PROCUREMENT Inclusion

* Any patient, regardless of age* or sex, with measurable EBV-positive Hodgkin's or non-Hodgkin's Lymphoma, (regardless of the histological subtype)^ or EBV (associated)- T/NK- or B cell lymphoproliferative disease

  * The first 3 patients enrolled will be adults. Patients <18 years of age are eligible if those first 3 patients do not experience dose limiting toxicity considered to be primarily related to the EBVST or Nivolumab.

  ^ Patients with relapsed or refractory lymphoma who failed or are ineligible for an autologous hematopoietic cell transplantation are also eligible for this study.
* EBV positive tumor (can be pending)
* Weighs at least 12kg
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given a copy of informed consent.
* Life expectancy of greater than 6 weeks.

TREATMENT Inclusion

- Any patient, regardless of age* or sex, with measurable EBV-positive Hodgkin's or non-Hodgkin's Lymphoma, (regardless of the histological subtype)^ or EBV (associated)-T/NK- or B cell lymphoproliferative disease

* The first 3 patients enrolled will be adults. Patients <18 years of age are eligible if those first 3 patients do not experience dose limiting toxicity considered to be primarily related to the EBVST or Nivolumab.

^ Patients with relapsed or refractory lymphoma who failed or are ineligible for an autologous hematopoietic cell transplantation are also eligible for this study.

And

* Hodgkin's lymphoma patients in second relapse or first relapse and refractory to at least two lines of salvage chemotherapy including Brentuximab Vedotin or primary refractory disease after at least two lines therapy or
* Non- Hodgkin's lymphoma patients in first relapse and/or refractory to at least one salvage chemotherapy or with primary refractory disease after at least two lines of therapy or in second or subsequent relapse or
* T/NK- or B lymphoproliferative disease in first relapse and/or refractory to at least one salvage chemotherapy or with primary refractory disease after at least two lines of therapy or in second or subsequent relapse
* EBV positive tumor
* Patients with life expectancy >/= 6 weeks.
* Patients with bilirubin less than or equal to 3x upper limit of normal
* AST less than or equal to 5x upper limit of normal
* Hgb more than 8.0 (may be a transfused value).
* Patients with a creatinine less than or equal to 2x upper limit of normal for age
* Pulse oximetry of more than 90% on room air
* Patients should have been off other investigational therapy for 4 weeks prior to entry in this study.
* Patients with a Karnofsky/Lansky score of >/= 60
* Recovered from acute toxic effects of prior chemotherapy at least one week before entering the study.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
* Informed consent explained to, understood and signed by patient/guardian. Patient/guardian given a copy of informed consent.

Exclusion Criteria:

PROCUREMENT Exclusion

* Active infection with HIV, HTLV, HBV, HCV (can be pending at this time)
* History of solid organ transplant

TREATMENT Exclusion

* Pregnant or lactating due to unknown effects of this therapy on a fetus or lactation
* Severe active intercurrent infection.
* Current use of systemic corticosteroids >0.5 mg/kg/day
* Currently receiving any investigational agents or radiotherapy within 4 weeks prior to entering the study.
* Patients with central nervous system involvement.
* History of allergic reactions attributed to nivolumab or any other checkpoint inhibitors.
* Uncontrolled autoimmune disease needing systemic steroids or steroid sparing agents except for hypothyroidism or type I diabetes.
* History of solid organ transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Lipase more than 70U/ml

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2020-07-11 (Actual)

PRIMARY OUTCOMES:
Number of Dose-Limiting Toxicities | 2 months
  For the purpose of this study, dose limiting toxicity will be defined as any of the below listed items considered to be primarily related to the EBVST infusion or Nivolumab:
  * CTCAE grade 3-4 diarrhea needing steroids for more than 1 week or needing hospitalization for more than 1 week,
  * Pancreatitis of any grade needing hospitalization,
  * Pneumonitis needing hospitalization for more than a week or needing home oxygen despite appropriate treatment for 1 week.
  * Hepatitis grade 3 or more not resolving in 2 weeks after discontinuation of therapy,
  * Stomatitis/mucositis needing TPN.
  * Musculoskeletal symptoms affecting activities of daily living for more than 2 weeks after discontinuation of therapy.

SECONDARY OUTCOMES:
Duration of Overall Response | Up to 1 year
  The duration of overall response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
  The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Pingali, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarathkumara YD, Van Bibber NW, Liu Z, Heslop HE, Rouce RH, Coghill AE, Rooney CM, Proietti C, Doolan DL. Differential antibody response to EBV proteome following EBVST immunotherapy in EBV-associated lymphomas. Blood Adv. 2025 Apr 8;9(7):1658-1669. doi: 10.1182/bloodadvances.2024014937. PMID 39908567

DOCUMENTS (1):
  • Informed Consent Form (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT02973113/ICF_000.pdf